CLINICAL TRIAL: NCT01248104
Title: Comparison of Tranexamic to Epsilon Aminocaproic Acid: a Prospective Analysis of Blood Conservation in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Jason Gatling, MD, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5100064
Record Dates: First submitted 2010-11-15; First posted 2010-11-25 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Cardiopulmonary Bypass
Keywords: Cardiac Surgery; Antifibrinolytic agents; Blood transfusion; epsilon aminocaproic acid; tranexamic acid
MeSH Terms: interventions — Tranexamic Acid; Aminocaproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Active Comparator): The research pharmacist used computer randomization to assign patients to receive either TXA or EACA. The TXA group re- ceived a bolus of 10 mg / kg over 15 minutes fol- lowed by an infusion of 1 mg/kg/hr.
  Interventions: Drug: Tranexamic Acid
- Aminocaproic Acid (Active Comparator): The research pharmacist used computer randomization to assign patients to receive either TXA or EACA. The EACA group received a bolus of 100 mg / kg given over 15 minutes shortly after induction of anesthesia followed by an infusion of 10 mg/kg/hr.
  Interventions: Drug: Aminocaproic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Infusion during cardiac surgery
  Other Names: TXA
  Arms: Tranexamic Acid
Drug: Aminocaproic Acid — Infusion during cardiac surgery
  Other Names: Amicar
  Arms: Aminocaproic Acid

SUMMARY:
We designed a prospective double-blinded randomized trial in an attempt to detect a difference between tranexamic acid (TXA) and epsilon aminocaproic acid (EACA) in reducing transfusion in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Background: This study compares the efficacy of tranexamic acid (TXA) to epsilon aminocaproic acid (EACA) in reducing blood loss in patients undergoing cardiac surgery. Methods: This was a double-blinded randomized trial. Patients (n=100) undergoing cardi- ac surgery were randomized to receive either TXA (10 mg/kg bolus followed by an infu- sion of 1mg/kg/hr) or EACA (150mg/kg bolus followed by an infusion of 20 mg/kg/hr). The primary outcome measure was a difference in transfusion amounts.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject 18 years of age or older?
2. Is the subject scheduled for primary cardiac surgery utilizing cardiopulmonary bypass(CPB)?
3. Is the subject more than 30 kg ( 66 lbs)?
4. Does subject understand English?

Exclusion Criteria:

1. Does the subject have existing coagulation defects (INR > 1.5, platelets < 100 ?
2. Does the subject have renal failure (defined as BUN/Cr ratio 20:1 ?
3. Does the subject have severe liver disease (AST & ALT> 3x normal) ?
4. Is the subject having emergency cardiac surgery, complex aortic surgery, combination valve/CABG surgeries, or redo cardiac surgery?
5. Is the subject having any procedure where CPB is not anticipated?
6. Is the patient weight greater than 150 kg?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gatling, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients scheduled for primary cardiac surgery utilizing CPB at LLUMC . Subjects myst be >30 kg, be able to understand English, and sign the consent form.Subjects will be recruited in the pre-admitting area prior to going to the PDCU area in the operating room.
Period: Overall Study
Arm/Group | Tranexamic Acid | Aminocaproic Acid
Started | 50 | 50
Completed | 40 | 42
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Aminocaproic Acid | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 38
  >=65 years | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.79175 (13.1260508) | 63.25333 (12.62622) | 63.51597561 (12.79547179)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 24 | 27 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Total Transfusion Amounts
Description: The outcome measure was the intergroup difference in total transfusion amounts up to post-operative day 2.
Time Frame: 48 hours
Population: equality in both arms
Measure: Mean (Standard Deviation); unit: mililiters
Arm/Group | Tranexamic Acid | Aminocaproic Acid
Number analyzed (Participants) | 40 | 42
mililiters | 161 (274) | 116 (296)
Statistical Analysis 1: Comparison: Tranexamic Acid vs Aminocaproic Acid; A power analysis based on the comparison of a 15% difference in total transfusion amounts up to POD 2 between the treatment groups indicated a total sample size of 80 with a power of 0.8, confidence interval 0.9, and p= 0.05; Test type: Superiority or Other — Continuous variables were compared by multivariate linear regression analysis to adjust for possible covariates of intraoperative fluids, age, bypass time, and procedure time. Tukey-Kramer test was then used to compare for specific differences between groups for each variable. Categorical data were compared using Fisher's exact test. All comparisons were made at a significance level of 0.05, and analysis was performed with Minitab version 17); p = 0.35, ANOVA — The primary outcome measure showed that there was no difference in PRBC transfusion frequency or amounts in the operating room or the in ICU up to POD 2

ADVERSE EVENTS:
Time Frame: length of hospital admission, an average of 5 days
Description: adverse events were recorded via review of electronic medical record
Arm/Group | Tranexamic Acid | Aminocaproic Acid
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes